CLINICAL TRIAL: NCT00436280
Title: An Open-label, Single Arm, Phase 2 Study of Rituximab, Gemcitabine and Oxaliplatin Plus Enzastaurin as Treatment for Patients With Relapsed Diffuse Large B-Cell Lymphoma
Brief Title: Chemotherapy for Participants With Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9819; H6Q-MC-S013 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Lymphoma, Large Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — enzastaurin; Gemcitabine; Rituximab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enzastaurin + Gemcitabine Rituximab Oxaliplatin (R-GEMOX) (Experimental)
  Interventions: Drug: enzastaurin; Drug: gemcitabine; Drug: rituximab; Drug: oxaliplatin

INTERVENTIONS:
Drug: enzastaurin — 1125 mg loading dose then 500 mg, oral, daily, until disease progression or 3 years
  Other Names: LY317615
Drug: gemcitabine — 1000 mg/m², IV, once, every two weeks, four to eight 2 week cycles
  Other Names: LY188011, Gemzar
Drug: rituximab — 375 mg/m², IV, once every 2 weeks, four to eight 2 week cycles
Drug: oxaliplatin — 100 mg/m², IV, once every two weeks, four to eight 2 week cycles

SUMMARY:
The primary purpose of this study is to help answer the following research questions:

* To assess whether Enzastaurin combined with rituximab, gemcitabine and oxaliplatin (R-GEMOX) can help participants with Diffuse Large B-Cell Lymphoma (DLBCL) remain free from disease and thus live longer.
* To assess for any side effects that might be associated with enzastaurin and R-GEMOX .
* To look at the characteristics and levels of certain genes and proteins to learn more about DLBCL and how enzastaurin works in the body.
* To look at the level of enzastaurin in the body and how long it remains.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DLBCL or transformed (cluster differentiation 20 [CD20]+) indolent lymphoma
* Relapsed/progressed after response obtained in 1st- or 2nd-line treatment, or participants who have not progressed after stable disease (SD) obtained in 1st- or 2nd-line.
* Measurable disease (lymph node greater than 1.5 cm)
* Adequate organ function
* Greater than or equal to 60 years or less than 60 (but greater than or equal to 18 years) who are not eligible for high-dose chemotherapy high-dose chemotherapy (HDC) and autologous stem cell transplant (ASCT)

Exclusion Criteria:

* Prior Allogeneic transplantation
* More than 2 prior anticancer treatment regimens
* Pregnant or breastfeeding
* Human-immunodeficiency-virus (HIV)associated lymphomas
* Brain metastases

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-02; Primary Completion 2009-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (18):
- France (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Créteil
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dijon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pessac
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pierre-Bénite
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rouen
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bremen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kassel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Reasons reported are for discontinuation from study treatment.
Groups:
- Enzastaurin + Gemcitabine Rituximab Oxaliplatin (R-GEMOX): Enzastaurin: 1125 milligram (mg) loading dose then 500 mg, orally, daily with Gemcitabine: 1000 milligram per square meter (mg/m²) administered intravenously (IV); Rituximab: 375 mg/m² IV; Oxaliplatin: 100 mg/m² IV all given once every 2 weeks (1 Cycle) for 4 Cycles for Induction. If responding participants receive 4 additional Cycles for consolidation, Enzastaurin will be given as maintenance until Progressive Disease (PD)/Toxicity or up to 3 years.
Period: Period 1: Induction
Arm/Group | Enzastaurin + Gemcitabine Rituximab Oxaliplatin (R-GEMOX)
Started | 68
Received at Least 1 Dose of Study Drug | 68
Completed | 40
Not Completed | 28
Not completed — Adverse Event | 8
Not completed — Progressive Disease | 12
Not completed — Stable Disease | 6
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Period: Period 2: Consolidation
Arm/Group | Enzastaurin + Gemcitabine Rituximab Oxaliplatin (R-GEMOX)
Started | 40
Completed | 23
Not Completed | 17
Not completed — Adverse Event | 1
Not completed — Progressive Disease | 10
Not completed — Stable Disease | 1
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 2
Not completed — Death | 1
Period: Period 3: Maintenance
Arm/Group | Enzastaurin + Gemcitabine Rituximab Oxaliplatin (R-GEMOX)
Started | 23
Completed | 5
Not Completed | 18
Not completed — Adverse Event | 6
Not completed — Progressive Disease | 12

BASELINE CHARACTERISTICS:
Groups:
- Enzastaurin + R-GEMOX: Enzastaurin: 1125 milligram (mg) loading dose then 500 mg, orally, daily with Gemcitabine: 1000 milligram per square meter (mg/m²) administered intravenously (IV); Rituximab: 375 mg/m² IV; Oxaliplatin: 100 mg/m² IV all given once every 2 weeks (1 Cycle) for 4 Cycles for Induction. If responding participants receive 4 additional Cycles for consolidation, Enzastaurin will be given as maintenance until Progressive Disease/Toxicity or up to 3 years.
Arm/Group | Enzastaurin + R-GEMOX
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.92 (12.468)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 68
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 68
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 10
  France | 41
  Germany | 17

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Progression Free Survival (PFS) After 1 Year Treatment
Description: PFS is defined as the rate at 1 year from the date of first dose of study drug to the first date of measured PD or death from any cause and was determined using the distribution of overall PFS times. The PFS rate at 1 year was determined using Kaplan-Meier estimates. For participants not known to have died as of the data cut-off date and who do not have PD, PFS was censored at the date of the last progression-free disease assessment.
Time Frame: First Dose of Study Drug to Measured Progressive Disease or Death from Any Cause at 1 Year
Population: All randomized participants who received at least 1 dose of study drug. Participants censored =14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin + R-GEMOX
Number analyzed (Participants) | 68
percentage of participants | 16.4 [8.1 to 27.4]

2. Secondary Outcome: Overall Response Rate (ORR) - Percentage of Participants Achieving Complete Response (CR) or Complete Response Unconfirmed (CRu) or Partial Response (PR) (Response)
Description: Assessment of response was based on the International Workshop to Standardize Response criteria for lymphoma (Cheson et al. 1999). CR is the complete disappearance of all detectable clinical and radiologic evidence of disease; all lymph nodes and nodal masses must have regressed to normal size (≤1.5 cm in their greatest transverse diameter for nodes >1.5 cm before therapy).CRu is as CR but with 1 or more of the following features: A residual lymph node mass >1.5 cm in greatest transverse diameter that has regressed by more than 75% in the sum of the products of the greatest diameters (SPD) and/or indeterminate bone marrow with normalization of all biologic abnormalities. PR is regression of more than 50% (SPD) of all measurable lesions, disappearance of nonmeasurable lesions and no new lesion. For each response category the number of participants with this response will be divided by the total number of participants treated to achieve the response rate.
Time Frame: Baseline to Measured Progressive Disease or Death from Any Cause at End of 4 and 8 Cycles
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin + R-GEMOX
Number analyzed (Participants) | 68
percentage of participants
  End of 4 cycles | 50 [37.60 to 62.40]
  End of 8 cycles: number analyzed (Participants) | 40
  End of 8 cycles | 52.50 [36.10 to 68.50]

3. Secondary Outcome: Percent of Participants With Progression-Free Survival (PFS) After 2 Years and 4 Years of Treatment
Description: PFS was defined as time from randomization until the first evidence of progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.0) or death from any cause; by Investigator assessment. Progressive disease (PD) was defined as at least a 20% increase in sum of longest diameter of target lesions taking as reference the smallest sum longest diameter since baseline, progression in non-target lesions or the appearance of 1 or more new lesion(s).
  PFS rate was defined as the rate of PFS at 2 year from the date of first dose of study drug and was determined using the distribution of overall PFS times.
  PFS rate was defined as the rate of PFS at 4 year from the date of first dose of study drug and was determined using the distribution of overall PFS times.
  For participants not known to have died as of the data cut-off date and who did not have PD, PFS was censored at the date of the last progression-free disease assessment.
Time Frame: First Dose of Study Drug to Measured Progressive Disease or Death from Any Cause at 2 Years, 4 Years
Population: All randomized participants who received at least 1 dose of study drug. 8 participants were censored.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin + R-GEMOX
Number analyzed (Participants) | 68
percentage of participants
  2 Years | 12.1 [5.5 to 21.6]
  4 Years | 8.7 [3.3 to 17.4]

4. Secondary Outcome: Percent of Participants With Overall Survival (OS) After 1 Year, 2 Years and 4 Years
Description: Overall survival was defined as the time from the date of first dose of study drug to the date of death from any cause. For participants who were not still alive at the time of analysis, survival time was censored at the last contact date. For participants not known to have died as of the cut-off date for analysis,OS was censored at the last contact date for participants in post-discontinuation.
Time Frame: First Dose of Study Drug to Death from Any Cause at 1 Year, 2 Years and 4 Years
Population: All randomized participants who received at least 1 dose of study drug. 14 participants were censored.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin + R-GEMOX
Number analyzed (Participants) | 68
percentage of participants
  1 Year | 52.3 [39.8 to 63.4]
  2 Years | 29.9 [19.5 to 41.0]
  4 Years | 20.9 [12.2 to 31.3]

5. Secondary Outcome: Percent of Participants With Event Free Survival (EFS) After 1 Year, 2 Years and 4 Years
Description: Event-free survival time was defined as the time from the date of first dose of study drug to the first date of measured PD,or start of a new treatment for the lymphoma, or death from any cause. For participants not known to have events as of the data cut-off date, EFS was censored at the date of the last tumor assessment.
Time Frame: First Dose of Study Drug to Measured PD, or Start of New Lymphoma Treatment or Death from Any Cause at 1 Year, 2 Years and 4 Years
Population: All randomized participants who received at least 1 dose of study drug. 6 participants were censored.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin + R-GEMOX
Number analyzed (Participants) | 68
percentage of participants
  1 Year | 15.0 [7.7 to 24.5]
  2 Years | 10.3 [4.4 to 19.0]
  4 Years | 8.6 [3.3 to 17.0]

6. Secondary Outcome: Progression-Free Survival (PFS ) of Participants With Diffuse Large B-cell Lymphoma (DLBCL) Germinal-Center B-cells (GCB) Versus Non-GCB Molecular Subtypes (Assessment of Biomarkers Relevant for Enzastaurin)
Description: PFS based on DLBCL molecular subtypes (GCB vs non-GCB) were determined. The molecular characterization of germinal center B-cells (GCBs) vs. non-GCBs was analyzed as separate combination immunohistochemistry (IHC) markers based on the Hans algorithms. Molecular subtype was included as class effect in the analytical models, adjusting for International Prognostic Index (IPI) score.
Time Frame: Baseline, Cycles 1-4, End of Study
Population: All randomized participants who received at least 1 dose of study drug and had evaluable samples.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin + R-GEMOX
Number analyzed (Participants) | 31
months
  GCB: number analyzed (Participants) | 10
  GCB | 7.8 [1.0 to 12.1]
  Non-GCB: number analyzed (Participants) | 21
  Non-GCB | 4.7 [2.0 to 7.3]
Statistical Analysis 1: Comparison: Enzastaurin + R-GEMOX; Comparing GCB versus non-GCB; Test type: Superiority or Other; Hazard Ratio (HR) = 0.512, 95% CI 2-sided [0.217 to 1.206] — Comparing GCB versus non-GCB

7. Secondary Outcome: PFS of Participants With Diffuse Large B-cell Lymphoma (DLBCL) Protein Kinase C Beta 2 (PKCB2) Expression (Assessment of Biomarkers Relevant for Enzastaurin)
Description: Reported PFS was based on PKCB2 protein expression assessed by immunohistochemistry (scored in 10% increments for percent of tumor cells). Protein expression levels was grouped into high and low in association with the clinical endpoints. Grouping was based on 1) a pre-specified threshold provided by the pathologist at Cleveland Clinic for the diffuse large B-cell lymphoma (DLBCL)-prognostic markers, and 2) a median cut-point for the enzastaurin-specific markers.
Time Frame: Baseline, Cycles 1-4, End of Study
Population: All randomized participants who received at least 1 dose of study drug and had evaluable samples.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin + R-GEMOX
Number analyzed (Participants) | 30
months
  High Expression: number analyzed (Participants) | 10
  High Expression | 3.6 [0.9 to 11.3]
  Low Expression: number analyzed (Participants) | 20
  Low Expression | 6.1 [1.8 to 7.9]
Statistical Analysis 1: Comparison: Enzastaurin + R-GEMOX; Comparing High Expression versus Low Expression; Test type: Superiority or Other; Hazard Ratio (HR) = 0.878, 95% CI 2-sided [0.388 to 1.989] — Comparing High Expression versus Low Expression

8. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration During a Dosing Interval at Steady State(Cmax,ss) for Total Analyte [Characterization of Pharmacokinetics of Enzastaurin and Its Metabolites]
Description: Cmax,ss is defined as the maximum observed drug concentration during a dosing interval at steady state. Non-Compartmental Pharmacokinetic Parameters for Total Analyte (Enzastaurin + LSN326020). LSN326020 is Enzastaurin's major active metabolite.
Time Frame: Day 2 of Cycle 2: Predose;1-2 Hours(H);3-4 h;5-6 h;7-8 H Postdose
Population: All randomized participants who received at least 1 dose of study drug and evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles per litre (nmol/L)
Arm/Group | Enzastaurin + R-GEMOX
Number analyzed (Participants) | 15
nanomoles per litre (nmol/L) | 2750 (61)

9. Secondary Outcome: PK: Area Under the Concentration vs. Time Curve During 1 Dosing Interval at Steady State (AUCτ,ss) for Total Analyte
Description: AUCτ,ss is defined as the area under the concentration versus time curve during 1 dosing interval at steady state.
Time Frame: Day 2 of Cycle 2: Predose;1-2 hours(h);3-4 h;5-6 h;7-8 h Postdose
Population: All randomized subjects who received at least 1 dose of study drug and evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles*hour per liter(nmol•h/L)
Arm/Group | Enzastaurin + R-GEMOX
Number analyzed (Participants) | 15
nanomoles*hour per liter(nmol•h/L) | 44100 (70)

10. Secondary Outcome: Percent of Participants With Disease-Free Survival (DFS) at 1 Year, 2 Years and 4 Years
Description: DFS was calculated as the duration from date of first dose of study drug to the date of first relapse event after CR or CRu or death from any cause. Participants who have not experienced an event at the time of analysis were censored at the most recent date of disease assessment. Events are relapse after a CR or CRu. Related death or death from unknown cause was considered as an event. Unrelated death was not considered as an event and the participant was censored at the time of death for this analysis. Unrelated death was defined as death from a cause not related to the lymphoma, any examination done for the lymphoma, or any treatment of the lymphoma.
Time Frame: First Dose of Study Drug to Relapse after CR or CRu or Death from any Cause at 1 Year, 2 Years and 4 Years
Population: All randomized participants who received at least 1 dose of study drug. 7 participants were censored.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin + R-GEMOX
Number analyzed (Participants) | 14
percentage of participants
  1 Year | 69.2 [37.3 to 87.2]
  2 Years | 52.7 [23.4 to 75.5]
  4 Years | 52.7 [23.4 to 75.5]

11. Secondary Outcome: Duration of Tumor Response (DOR)
Description: Duration of tumor response was defined as the time from the date when the measurement criteria were met for CR and CRu or PR (whichever status was recorded first) until the date of first observation of objective disease progression. For responding patients who died without objective PD (including death from study disease), duration of response was censored at the date of the last objective progression-free disease assessment. For responding patients not known to have died as of the data cut-off date and who do not have objective PD, duration of response was censored at the date of the last objective progression-free disease assessment. For responding patients who received subsequent systemic anticancer therapy (after discontinuation from the study chemotherapy) prior to objectively determined disease progression, duration of response was censored at the date of the last objective progression-free disease assessment prior to post-discontinuation therapy.
Time Frame: Time from Observed CR and CRu or PR (Up to 4 Years)
Population: All randomized participants who received at least 1 dose of study drug. Participants censored =13.
Measure: Number (95% Confidence Interval); unit: years
Arm/Group | Enzastaurin + R-GEMOX
Number analyzed (Participants) | 3
years | 23.4 [9.6 to 40.6]

ADVERSE EVENTS:
Groups:
- Enzastaurin + R-GEMOX: enzastaurin: 1125 mg loading dose then 500 mg, oral, daily, until disease progression or 3 years
  gemcitabine: 1000 mg/m2, IV, once, every two weeks, four to eight 2 week cycles
  rituximab: 375 mg/m2, IV, once every 2 weeks, four to eight 2 week cycles
  oxaliplatin: 100 mg/m2, IV, once every two weeks, four to eight 2 week cycles
Arm/Group | Enzastaurin + R-GEMOX
Serious Adverse Events (participants affected / at risk) | 30/68
Other Adverse Events (participants affected / at risk) | 68/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Enzastaurin + R-GEMOX (N=68)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (4)
Atrial flutter (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Jejunitis (Gastrointestinal disorders) | 1 (2)
Death (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (3)
General physical health deterioration (General disorders) | 2 (9)
Pyrexia (General disorders) | 5 (7)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (3)
Septic shock (Infections and infestations) | 1 (2)
Tooth abscess (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (11)
Upper respiratory tract infection (Infections and infestations) | 1 (2)
Viral infection (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (3)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (6)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/21 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (2)
Dysaesthesia (Nervous system disorders) | 1 (8)
Hypogeusia (Nervous system disorders) | 1 (8)
Haematuria (Renal and urinary disorders) | 1 (2)
Renal cyst haemorrhage (Renal and urinary disorders) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (2)
Urinary retention (Renal and urinary disorders) | 1 (4)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Thrombophlebitis (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin + R-GEMOX (N=68)
Anaemia (Blood and lymphatic system disorders) | 34 (115)
Leukopenia (Blood and lymphatic system disorders) | 34 (109)
Lymphopenia (Blood and lymphatic system disorders) | 25 (75)
Neutropenia (Blood and lymphatic system disorders) | 42 (151)
Thrombocytopenia (Blood and lymphatic system disorders) | 44 (188)
Abdominal pain (Gastrointestinal disorders) | 7 (12)
Constipation (Gastrointestinal disorders) | 13 (41)
Diarrhoea (Gastrointestinal disorders) | 19 (40)
Nausea (Gastrointestinal disorders) | 26 (58)
Vomiting (Gastrointestinal disorders) | 14 (23)
Asthenia (General disorders) | 16 (51)
Fatigue (General disorders) | 9 (30)
Mucosal inflammation (General disorders) | 4 (5)
Oedema peripheral (General disorders) | 10 (15)
Pyrexia (General disorders) | 9 (14)
Urinary tract infection (Infections and infestations) | 5 (8)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (5)
Alanine aminotransferase increased (Investigations) | 21 (59)
Aspartate aminotransferase increased (Investigations) | 22 (74)
Blood creatinine increased (Investigations) | 4 (17)
Blood lactate dehydrogenase increased (Investigations) | 12 (42)
Weight decreased (Investigations) | 8 (22)
Decreased appetite (Metabolism and nutrition disorders) | 7 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (9)
Neuropathy peripheral (Nervous system disorders) | 8 (40)
Paraesthesia (Nervous system disorders) | 19 (97)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (60)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days